CLINICAL TRIAL: NCT04443101
Title: Comparison of Changes in Effective Lens Position of Different Types of Intraocular Lens
Brief Title: Effective Lens Position After Cataract Surgery
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Wenzhou Medical University (Other)
Responsible Party: Principal Investigator, yin ying zhao, Principal Investigator, Wenzhou Medical University
Other Study IDs: SSOCT-ELP
Record Dates: First submitted 2020-06-17; First posted 2020-06-23 (Actual); Last update posted 2023-03-07 (Actual); Status verified 2023-03

CONDITIONS: Age-related Cataract

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group（SN6CWS）: Group（SN6CWS）：Implant SN6CWS intraocular lens
  Interventions: Other: different types of intracular lens
- Group（MI60）: Group（MI60）：Implant MI60 intraocular lens
  Interventions: Other: different types of intracular lens
- Group（Aspira-aA）: Group（Aspira-aA）：Implant Aspira-aA intraocular lens
  Interventions: Other: different types of intracular lens

INTERVENTIONS:
Other: different types of intracular lens — different types of intracular lens

SUMMARY:
Cataract patients were implanted with different types of intraocular lenses for grouping. SSOCT scanning was used to measure ELP and optometry.

DETAILED DESCRIPTION:
Cataract patients were implanted with different types of intraocular lenses for grouping. Perform SSOCT scan that was used to measure effective lens position and optometry at different postoperative follow-up time .

ELIGIBILITY:
Inclusion Criteria:

* a.Diagnosed as cataract;
* b.Implanted intraocular lens: SN6CWS, Aspira-aA, MI60;
* c.Cataract phacoemulsification and intraocular lens implantation.

Exclusion Criteria:

* a.Combined with corneal opacity, glaucoma, uveitis, retinal detachment and other eye diseases;
* b.A history of intraocular surgery or trauma other than cataract surgery;
* c.Intraoperative complications such as tearing of the capsule and IOL failure to implant;
* d.Endophthalmitis, corneal endothelial decompensation and other postoperative complications;
* e.Those with incomplete data collected during the follow-up period of postoperative patients.

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * Diagnosed as cataract in our hospital;
  * Implanted intraocular lens: SN6CWS, Aspira-aA, MI60;
  * Cataract phacoemulsification and intraocular lens implantation.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2022-05-30 (Actual); Study Completion 2023-03-30 (Estimated)

PRIMARY OUTCOMES:
effective lens position | up to 3 months after cataract surgery
  Changes of effective lens position at different time points after cataract surgery

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Ophthalmology and Optometry Hospital, Wenzhou, Zhejiang
  - Wenzhou Medical University, Wenzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No